CLINICAL TRIAL: NCT06624878
Title: Intraoperative Esketamine for Prevention of Depressive Symptoms After Cytoreductive Surgery in Ovarian Cancer: a Controlled, Randomized Clinical Trial
Brief Title: Esketamine for Prevention of Depression After Cytoreductive Surgery in Ovarian Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Gu Bin, Clinical Professor, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-2024-885 (IIT)
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-10

CONDITIONS: Ovarian Cancer; Cytoreductive Surgery; Depressive Symptom
MeSH Terms: conditions — Ovarian Neoplasms; Depression | interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the esketamine group (Experimental)
  Interventions: Drug: esketamine
- the placebo group (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: esketamine — 0.2 mg/kg esketamine infused intravenously after induction of general anesthesia.
  Arms: the esketamine group
Drug: placebo — a placebo (an equivalent volume of normal saline) infused intravenously after induction of general anesthesia.
  Arms: the placebo group

SUMMARY:
The goal of this clinical trial is to learn if intraoperative administration of esketamine would prevent or mitigate postoperative depressive symptoms after cytoreductive surgery in ovarian cancer. The main questions it aims to answer are:

* Whether a single low dose of esketamine administered would reduce the postoperative depressive symptoms three days after cytoreductive surgery in ovarian cancer?
* Whether a single low dose of esketamine administered would relief the postoperative sleep disturbance, postoperative recovery? Researchers will compare the esketamine to a placebo (normal saline) to see if the esketamine works to reduce the postoperative depressive symptoms.

Participants will:

* Receive either 0.2 mg/kg esketamine or placebo infused intravenously after induction of general anesthesia.
* The preoperative Patient Health Questionnaire 9 (PHQ-9) scale was used to verify the symptoms suggestive of depression.

ELIGIBILITY:
Inclusion Criteria:

* undergoing cytoreductive surgery for ovarian cancer under general anesthesia
* ASA physical status I-III
* Ages 18-80 years

Exclusion Criteria:

* Patients taking anti-psychotic medications
* Contraindications to esketamine
* Language barrier
* Inability to provide consent

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of postoperative depressive symptoms after cytoreductive surgery in ovarian cancer | on postoperative day 3
  The postoperative depressive symptoms are assessed using the preoperative Patient Health Questionnaire 9 (PHQ-9) scale. The range of this scale is 0-27, and a standard threshold score of 10 or higher indicates symptoms of depression.

SECONDARY OUTCOMES:
the incidence of depressive symptoms in ovarian cancer | Baseline (before surgery), on postoperative day 30
  The PHQ-9 was also used to assess the depressive symptoms.The range of this scale is 0-27, and a standard threshold score of 10 or higher indicates symptoms of depression.
the incidence of sleep disturbance in ovarian cancer | Baseline (before surgery), on postoperative day 3 and on postoperative day 30
  The sleep disturbance are assessed using the Athens Insomnia Scale (AIS). The range of this scale is 0-24, and a standard threshold score of 7 or higher indicates sleep disturbance.
the incidence of anxiety in ovarian cancer | Baseline (before surgery)
  The anxiety symptom is assessed using the Generalized Anxiety Disorder-7 (GAD-7). The range of this scale is 0-21, and a standard threshold score of 10 or higher indicates anxiety.
the postoperative recovery of ovarian cancer | Baseline (before surgery), on postoperative day 3
  The postoperative recovery is assessed using the quality of recovery-15 questionnaire (QoR-15) .The QoR-15 has 15 questions. Each question is rated on a 10-point scale, ranging from 0 (none of the time or poor) to 10 (all of the time or excellent). The maximum score (best recovery) is 150.
postoperative pain score at rest and coughing pain | at 1, 24, 48, 72 hours after surgery
  The postoperative pain at rest and during coughing are assessed by NRS score with a range of 0 to 10 (0=no pain, 10=the worst possible pain).
the lengh of postoperative ICU admission | through study completion, an average of 1-5 days
the time to initiation of postoperative chemotherapy | through study completion, an average of 5-20 days
the postoperative complications of ovarian cancer | within 30 days after surgery
  The complications are assessed using the Claviene-Dindo score.
the time to walk after surgery | through study completion, an average of 2-5 days
the time to return of bowel function | through study completion, an average of 5-10 days
the time to readiness for discharge | through study completion, an average of 7-15 days
morphine requirements after surgery | at 24 hours after surgery
morphine requirements after surgery | at 48 hours after surgery
the residual disease after cytoreductive surgery | on postoperative day 1
  The residual disease is assessed using the propotion of optimal debulking.
the incidence of nausea and vomiting | during 72 hours after surgery
the incidence of postoperative hypotension | during 72 hours after surgery
the incidence of pruritus | during 72 hours after surgery
the incidence of drowsiness | during 72 hours after surgery
the incidence of respiratory depression | during 72 hours after surgery
the incidence of nystagmus | during 72 hours after surgery
the incidence of diplopia | during 72 hours after surgery
the incidence of hypertonia | during 72 hours after surgery
the incidence of daymare | during 72 hours after surgery
the incedence of neuropsychiatric symptoms | during 72 hours after surgery
  The neuropsychiatric symptoms are assessed using BPRS-4. The range of this scale is 0-28, and a standard threshold score of 5 or higher indicates symptoms of neuropsychiatric symptoms.
the incidence of dissociative states | during 72 hours after surgery
  The dissociative states are assessed using the CADSS-6. The range of this scale is 0-24, and a standard threshold score of 3 or higher indicates symptoms of dissociative states.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang cancer hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
We will share data on ClinicalTrials.gov, and data sharing will be always available.
Supporting Information: Study Protocol, SAP
Time Frame: starting about 6 months after publication